CLINICAL TRIAL: NCT04777240
Title: Characterization of Enterococci; Distribution of Virulence Markers, Virulence Genes and Antibiotic Resistance Pattern of the Isolated Species
Brief Title: Characterization of Enterococci
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ekram Abd El Rahman Mahmoud, Medical Microbiology Department, faculty of Medicine, Sohag University
Other Study IDs: Soh-Med-21-02-19
Record Dates: First submitted 2021-02-20; First posted 2021-03-02 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-02

CONDITIONS: Samples From Patients With Enterococcal Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study on Characterization of Enterococci because nowadays it become an important cause of nosocomial infections .detection of the most common two species of Enterococci and most common virulence factors & its genes with determination of antibiotics sensitivity test for the isolated strains

ELIGIBILITY:
Inclusion Criteria:

* any patients in ICU has manifestations of urinary tract infections, surgical wound infections, intra-abdominal infections, intrapelvic infections, bacteraemia and infective endocarditis

Exclusion Criteria:

* patients receiving antibiotics in previous 48 hours

Ages: 2 Months to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients in ICU in Sohag University Hospital
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
I) Sample collection | 2 months
  Samples are collected from intensive care unit (ICU) including urine, pus swabs, sputum, blood, tracheal aspirates and pharyngeal swabs
II) Identification of Enterococci: | 2 month
  by inoculation on Bile esculin azide & growing colonies further identified by :
  1. microscopically after staining by gram stain
  2. catalase test
  3. grow on high concentration of NaCl (6.5%)
III) Phenotypic detection of virulence marker of Enterococci(Gelatinase activity) | 2 weeks
  by culture on nutrient agar containing gelatin.Positive results appeared as liquefaction of gelatin
IV)Phenotypic detection of virulence marker of Enterococci (hemolytic activity) | 1 week
  by Detection of hemolytic activity on the blood agar
V) Phenotypic detection of virulence marker of Enterococci(Caseinase production) | 2 weeks
  by Detection of Caseinase production on Muller hinton agar containing skimmed milk 3%.
VI) Phenotypic detection of virulence marker of Enterococci(Formation of Slime layer) | 1 week
  Formation of Slime layer by culture on Brain heart infusion agar containing 5% sucrose, plates are incubated for 24 hrs at 37oC. Positive strains gave mucoid and slimy colonies.
VII) Phenotypic detection of virulence marker of EnterococcI (Biofilm formation) | 2 weeks
  using microtiter plate reader. Biofilm formation is scored as nonbiofilm forming (-), weak - (+), moderate - (++), and strong - (+++) corresponding to the A630 values ≤1, 1-≤2, 2-≤3, and>3, respectively
VIII) Antibiotic sensitivity test: | 3 monthe
  1. by 1- disc diffusion test using Vancomycin 30 μg, Teichoplanin 30 μg, Tetracycline 30 μg, Ampicillin 10 μg and Erythromycin 15 μg. Results ,Results are interpreted according to CLSI 2018.
  2. E-test:
  MICs (minimal inhibitory concentrations) of Vancomycin are measured by E-test for confirmation of vancomycin resistance among the isolated Enterococci. Results are interpreted according to CLSI guidelines.
IX) Molecular Identification of commonest Enterococcus species | 1 month
  by conventional gene specific uniplex PCR for E. faecalis and E. Faecium
X) Molecular detection of virulence genes | 2 months
  Identification of virulence genes; gel E (gene for gelatinase), asa1 (gene for aggregation substance), cylA (gene for cytolysin activator), esp (gene for Enterococcal surface protein) Hyl (gene for Hyaluronidase) of E. faecalis and E. faecium was performed by uniplex PCR.The amplified products are visualized on 2% agarose gel stained with ethidium bromide. The stained gels are visualized and documented with a gel documentation system and analyzed visually to determine the size of PCR amplicons of the target genes directly by comparison with 100 bp DNA ladder marker.

CONTACTS AND LOCATIONS:
Overall Officials: Ekram Ab Rahmand Mahmoud, lecturer, Principal Investigator — Sohag Faculty of Medicine
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No